CLINICAL TRIAL: NCT00983944
Title: A Randomized Phase II Study of Dose-Adjusted EPOCH-R and R-VACOP-B in Primary Mediastinal (Thymic) Large B-Cell Lymphoma
Brief Title: Rituximab and Combination Chemotherapy With or Without Bleomycin Sulfate in Treating Patients With Primary Mediastinal Large B-Cell Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate Accrual
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-08178; NCI-2011-03123 (Registry Identifier: Clinical Trial Reporting Program (CTRP))
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Lymphoma
Keywords: contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; childhood diffuse large cell lymphoma; stage I childhood large cell lymphoma; stage II childhood large cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Dendritic Cell Sarcoma, Interdigitating | interventions — Bleomycin; Rituximab; EPOCH protocol; Cyclophosphamide; Doxorubicin; Etoposide; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (EPOCH-R) (Experimental): Patients receive rituximab IV on day 1; etoposide IV, doxorubicin hydrochloride IV, and vincristine sulfate IV continuously over 96 hours on days 1-4; cyclophosphamide IV over 30 minutes on day 5; and oral prednisone twice daily on days 1-5. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: rituximab; Drug: EPOCH regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: prednisone; Drug: vincristine sulfate
- Arm II (R-VACOP-B) (Experimental): Patients receive rituximab IV and doxorubicin hydrochloride IV on day 1 of weeks 1, 3, 5, 7, 9, and 11; cyclophosphamide IV over 30 minutes on day 1 of weeks 1, 5, and 9; etoposide IV over 1 hour on day 1 and then orally on days 2 and 3 of weeks 3, 7, and 11; bleomycin sulfate IV and vincristine sulfate IV on day 1 of weeks 2, 4, 6, 8, 10, and 12; and oral prednisone on days 1-7 of week 1 and then every other day in weeks 2-10.
  Interventions: Biological: bleomycin sulfate; Biological: rituximab; Drug: EPOCH regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: prednisone; Drug: vincristine sulfate

INTERVENTIONS:
Biological: bleomycin sulfate — Given IV
  Arms: Arm II (R-VACOP-B)
Biological: rituximab — Given IV
Drug: EPOCH regimen — Given IV or orally
Drug: cyclophosphamide — Given IV or orally
Drug: doxorubicin hydrochloride — Given IV or orally
Drug: etoposide — Given IV or orally
Drug: prednisone — Given IV or orally
Drug: vincristine sulfate — Given IV or orally

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving rituximab together with combination chemotherapy may kill more cancer cells. It is not yet known which combination chemotherapy regimen is more effective when given with rituximab in treating large B-cell lymphoma.

PURPOSE: This randomized phase II trial is studying how well rituximab and combination chemotherapy work when given with or without bleomycin sulfate in treating patients with primary mediastinal large B-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the complete response rate based on PET/CT scan criteria in patients with primary mediastinal large B-cell lymphoma (PMLCL) treated with dose-adjusted rituximab, etoposide, doxorubicin hydrochloride, vincristine sulfate, cyclophosphamide, and prednisone with or without bleomycin sulfate.

Secondary

* To characterize the progression-free survival (PFS) of patients treated with these regimens.
* To assess the toxicity profiles associated with these regimens in these patients.
* To determine the prognostic significance of a mid-therapy PET scan and an end-of-therapy PET scan in achieving complete response and in predicting 2-year PFS of patients treated with these regimens.
* To explore the effect of involved-field radiotherapy on 2-year PFS of patients who are PET positive at the end of chemotherapy.
* To explore the efficacy of an end-of-therapy PET/CT scan in predicting which patients can avoid radiotherapy.
* To characterize the overall survival of patients treated with these regimens.
* To prospectively validate a pattern of immunohistochemical staining, including nuclear c-REL, TRAF-1, c-JUN, and Gal1, to accurately distinguish PMLCL from other lymphoid malignancies.
* To determine if levels of soluble CD30 correlate with disease activity in PMLCL.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I (EPOCH-R): Patients receive rituximab IV on day 1; etoposide IV, doxorubicin hydrochloride IV, and vincristine sulfate IV continuously over 96 hours on days 1-4; cyclophosphamide IV over 30 minutes on day 5; and oral prednisone twice daily on days 1-5. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
* Arm II (R-VACOP-B): Patients receive rituximab IV and doxorubicin hydrochloride IV on day 1 of weeks 1, 3, 5, 7, 9, and 11; cyclophosphamide IV over 30 minutes on day 1 of weeks 1, 5, and 9; etoposide IV over 1 hour on day 1 and then orally on days 2 and 3 of weeks 3, 7, and 11; bleomycin sulfate IV and vincristine sulfate IV on day 1 of weeks 2, 4, 6, 8, 10, and 12; and oral prednisone on days 1-7 of week 1 and then every other day in weeks 2-10.

In both arms, patients undergo PET/CT scans at baseline, mid-therapy, and after completion of chemotherapy. Patients with stable or progressive disease after completion of chemotherapy are removed from the study. Patients with complete response undergo observation. Patients with partial response undergo involved-field radiotherapy to any area of bulky disease at diagnosis and to any FDG-avid area on PET scan 3-4 weeks after completion of chemotherapy. These patients then undergo additional PET/CT scan at 8-10 weeks after completion of radiotherapy.

Blood samples are collected at baseline, during mid-therapy restaging, and after completion of chemotherapy for analysis of soluble CD30 levels by ELISA. Previously collected tissue samples are obtained for biomarker analysis by IHC.

After completion of study therapy, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary mediastinal (thymic) large B-cell lymphoma as defined by WHO classification of lymphoid neoplasms

  * Diagnosis must be based on an adequate tissue sample, such as an excisional biopsy or core-needle biopsy
* A paraffin-embedded block of well-fixed lymphoma tissue must be available
* Measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension as ≥ 10 mm
* No active or untreated CNS lymphoma

  * A lumbar puncture is not required in the absence of neurologic symptoms

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* ANC ≥ 1,000/mm^3 (unless related to disease)
* Platelet count ≥ 100,000/mm^3 (unless related to disease)
* Total bilirubin ≤ 2.0 times upper limit of normal (ULN)
* AST and/or ALT ≤ 2.5 times ULN
* Creatinine ≤ 2.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Ejection fraction ≥ 45% by MUGA or echocardiogram
* Patients with HIV infection are eligible, provided the following criteria are met:

  * No evidence of co-infection with hepatitis B or C
  * CD4 cell count ≥ 400/mm^3
  * No evidence of resistant strains of HIV
  * HIV viral load ≤ 10,000 copies HIV RNA/mL (if not on anti-HIV therapy)
  * HIV viral load ≤ 50 copies HIV RNA/mL (if on anti-HIV therapy)
  * No history of AIDS-defining conditions
* No concurrent uncontrolled illness including, but not limited to, the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situation that would limit compliance with study requirements
* No active secondary malignancy except nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY:

* No prior cytotoxic chemotherapy or rituximab

  * Prior limited course of glucocorticoids allowed
* No other concurrent investigational or commercial anticancer therapies

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2011-04-25 (Actual); Study Completion 2011-04-25 (Actual)

PRIMARY OUTCOMES:
Complete response rate | Up to a year

SECONDARY OUTCOMES:
Two-year progression-free survival | Up to 2 years
Overall survival | Up to 3 years
Toxicity as assessed by NCI CTCAE v3.0 | Up to 3 years
Immunohistochemical staining results | Up to a year
Correlation of soluble CD30 levels with disease activity in PMLCL | Up to a year

CONTACTS AND LOCATIONS:
Overall Officials: Kristie A. Blum, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center